CLINICAL TRIAL: NCT06674655
Title: Motor Imagery and Therapeutic Exercise on Sensorimotor Function in Women With Menstrual Pain: A Randomized Controlled Trial
Brief Title: Motor Imagery Plus Therapeutic Exercise in Women With Menstrual Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Ferran Cuenca, Doctor of Physical Therapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UV0004
Record Dates: First submitted 2024-11-02; First posted 2024-11-05 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Motor Imagery Training
Keywords: Motor Imagery; Therapeutic Exercise; Menstrual Pain
MeSH Terms: conditions — Dysmenorrhea | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor Imagery Plus Therapeutic Exercise (Experimental)
  Interventions: Behavioral: Motor Imagery Plus Therapeutic Exercise
- Therapeutic Exercise (Active Comparator)
  Interventions: Behavioral: Therapeutic Exercise
- Minimal Intervention (Sham Comparator)
  Interventions: Behavioral: Minimal intervention

INTERVENTIONS:
Behavioral: Motor Imagery Plus Therapeutic Exercise — This group will perform three days of lumbo-pelvic motor control exercise intervention along with a motor imagery intervention program during active breaks between exercises.
  Arms: Motor Imagery Plus Therapeutic Exercise
Behavioral: Therapeutic Exercise — This group will perform a lumbo-pelvic motor control exercise program for three consecutive days.
  Arms: Therapeutic Exercise
Behavioral: Minimal intervention — This group will carry out a therapeutic counseling and minimal education intervention during a one-day intervention.
  Arms: Minimal Intervention

SUMMARY:
The researchers will conduct a study that combines motor imagery with therapeutic exercise in women experiencing menstrual pain. Previous research suggests that motor imagery, when used alongside physical exercise, may help improve motor control and alleviate pain, potentially enhancing outcomes for individuals dealing with chronic pain conditions. Through this study, the investigators aim to explore the effectiveness of these interventions in targeting key variables such as pain perception, motor coordination, and overall quality of life, building on existing evidence of motor imagery's benefits in pain management.

ELIGIBILITY:
Inclusion Criteria:

* Women who have experienced menstrual pain for more than 6 months.
* Pain intensity rated higher than 3/10 on a pain scale.
* Participants do not take pain-relief medication during the study period.
* Ages between 18 and 35 years old

Exclusion Criteria:

* Current use of hormonal contraceptives or other treatments that affect menstrual cycles.
* Any chronic pain condition unrelated to menstrual pain (e.g., fibromyalgia, chronic low back pain).
* Diagnosed gynecological conditions such as endometriosis or pelvic inflammatory disease.
* Pregnancy or breastfeeding.
* Current use of psychoactive medications that could affect pain perception.
* Any significant psychiatric condition that could interfere with study participation.
* History of recent pelvic surgery (within the last 6 months).

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-01-09 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Menstrual pain intensity will be assessed pre-intervention (T0), mid-intervention (T1-day 1, T2-day 2) and Post-intervention (T3-day 3).
  The main variable is the intensity of menstrual pain, which will be evaluated before, during and after the intervention using a verbal numerical scale (0-10), where 0 is no pain and 10 is maximum pain.

SECONDARY OUTCOMES:
Lumbopelvic Motor Control | Lumbopelvic motor control will be assessed pre-intervention (T0), mid-intervention (T1-day 1, T2-day 2) and Post-intervention (T3-day 3).
  Lumbopelvic motor control will be assessed by a visual feedback system starting from a pressure of 40 mmHg.
Pain Sensitivity | Pain sensitivity will be assessed pre-intervention (T0), mid-intervention (T1-day 1, T2-day 2) and Post-intervention (T3-day 3).
  Pain sensitivity will be assessed with an algometer using pressure pain thresholds (in various areas, such as the abdomen, lumbar and thiabial region), as well as through conditioned pain modulation.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valènica, Spain